CLINICAL TRIAL: NCT02907151
Title: Evaluation of the Contribution of a Pre-consultation Questionnaire on the Therapeutic Education of Patients on Anticoagulants During a Routine Inspection by the Cardiologist.
Brief Title: Evaluation of the Contribution of a Pre-consultation Questionnaire on the Therapeutic Education
Acronym: EDUCONSULT
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL16_0275
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2016-09

CONDITIONS: Under Oral Anticoagulation Patients
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- pre-consultation survey group: The group completing a pre consultation survey filled the same questionnaire in post consultation but the doctor will see the result in the consultation.
  Interventions: Other: Survey
- Group absence of pre-consultation survey: This group will be a control group to see if there is a difference between completing a pre-consultation survey before or not.

INTERVENTIONS:
Other: Survey — Complete a survey prior to the consultation and a questionnaire after
  Groups: pre-consultation survey group

SUMMARY:
To assess the value of a dedicated knowledge questionnaire, filled by the patient prior consultation. Indeed, it could allow to target specific shortcomings of patients first, and help the cardiologist to prioritize the other therapeutic education, targeting specifically the information provided.

DETAILED DESCRIPTION:
The main objective is to study the impact of a pre-consultation questionnaire on the knowledge gained by the patient on anticoagulant treatment at the exit of cardiology consultation.

The assumption is that this questionnaire would help educate patients about their shortcomings and educate cardiologists lack of knowledge of his patient.

The secondary objectives are :

* Target specific areas in which patients have the greatest lack of information
* Assess the impact of educational level on information
* Assess the impact of age on information
* Evaluate the satisfaction of the information delivered
* Assess patient anxiety vis-à-vis their treatment
* Evaluate the failure rate of the questionnaire to know the number of patients refusing to participate in the study

ELIGIBILITY:
Inclusion Criteria:

* Patient monitoring Cardiology Consultation at University Hospital of Montpellier, whatever the reason
* Patients on oral anticoagulant therapy (warfarin or AOD) for over a month.

Exclusion Criteria:

* Severe cognitive disorders, making it impossible to understand the patient on therapeutic education.
* Disorders of the important vision.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for cardiac consultation treated with oral anticoagulation
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
number of correct answers | 3 months
  score (number of correct answers) to the survey

SECONDARY OUTCOMES:
Score information | 3 months
  Score information for the different areas of the survey
Score on the provision of additional information | 3 months
  Score on the provision of additional information in the consultation.
anxiety score | 3 months
  anxiety score by a self-evaluation of the patient.
Score information based on subgroups | 3 months
  Score information based on subgroups:
  * level of education
  * Age
  * Sex

CONTACTS AND LOCATIONS:
Overall Officials: Florence Leclercq, MD PHD, Study Director — University Hospital, Montpellier
Locations (1):
- Leclercq, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided